CLINICAL TRIAL: NCT05707845
Title: Effect of Weight Reduction and Aerobic Exercise on Premenstrual Syndrome Symptoms in Obese Females
Brief Title: Effect of Weight Reduction and Aerobic Exercise on PMS Symptoms in Obese Females
Acronym: PMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yara Mostafa Soliman Mahmoud Abdlbary, M.SC physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 012/003813
Record Dates: First submitted 2023-01-08; First posted 2023-02-01 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Premenstrual Syndrome
Keywords: "premenstrual syndrome"; "diet"; "exercise"; "obesity"
MeSH Terms: conditions — Premenstrual Syndrome; Motor Activity; Obesity | interventions — Anti-Inflammatory Agents, Non-Steroidal; Exercise

STUDY DESIGN:
Intervention Model Description: * Two groups pre-test post-test design.
  * In this study the patients will be randomly assigned into two equal groups (20 patients for each group).
    (a) Group A: (control group):
  * Medical treatment in the form of nonsteroidal anti-inflammatory drugs (NSAIDs). (b) Group B: (Study group):
  * Medical treatment in the form of nonsteroidal anti-inflammatory drugs (NSAIDs).
  * Physical therapy program weight reduction by diet program in the form of caloric restriction, in combination to aerobic exercise in the form of using treadmill 30 minutes /3 times a week for 12 weeks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (A) (Placebo Comparator): Group A: (control group): 20 participants Medical treatment in the form of nonsteroidal anti-inflammatory drugs (NSAIDs)
  Interventions: Drug: Medical treatment.
- study group (B) (Experimental): Group B: (Study group): 20 participants
  * Medical treatment in the form of nonsteroidal anti-inflammatory drugs (NSAIDs).
  * Physical therapy program weight reduction by diet program in the form of caloric restriction, in combination to aerobic exercise in the form of using treadmill 30 minutes /3 times a week for 12 weeks.
  Interventions: Drug: Medical treatment.; Behavioral: weight reduction; Other: exercise

INTERVENTIONS:
Drug: Medical treatment. — Medical treatment in the form of nonsteroidal anti-inflammatory drugs (NSAIDs).
  Other Names: NSAID
Behavioral: weight reduction — weight reduction in the form low caloric diet program for 12 weeks.
  Other Names: diet program
  Arms: study group (B)
Other: exercise — aerobic exercise in the form of walking on treadmill for 30 minutes 3 times a week for 12 weeks.
  Other Names: aerobic exercise
  Arms: study group (B)

SUMMARY:
The purpose of this study will be investigation of the effect of weight reduction and aerobic exercises on premenstrual syndrome symptoms in obese females.

DETAILED DESCRIPTION:
both groups (A&B) will take their medical treatment in the form of (NSAIDs) and the study group B will under go a siet plan which will fits the participants. Diet plan extends for 12 weeks in the form of caloric restriction program and each woman in group B will perform aerobic exercise program, in the form of treadmill 3 times/week for 8 weeks for 12 weeks. Each session will take about 30 minutes as the following: 5 minutes warming up exercises by walking on the treadmill by low speed, 20 minutes walking at moderate intensity (70% of the maximal heart rate) and 5 minutes are cooling down by walking on the treadmill by low speed as in warming up.

ELIGIBILITY:
Inclusion Criteria:

* Age will range between 20- 30 years old.
* only females will participate in the study.
* All patients who will be enrolled to the study will have their informed consent.

Exclusion Criteria:

* Diabetes mellitus.
* Individuals with cardiopulmonary conditions.
* Individuals with any pelvic disease.
* Individuals undergoing radiation therapy or chemotherapy.
* Hepatic or pancreatic diseases.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — females
Enrollment: 40 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Progesterone levels in blood | 12 weeks
  progesterone level will be checked six to eight days after ovulation start (about day 21st of a 28-day cycle)
body weight | 12 weeks
  Weight and height measurement will be measured while the woman is wearing a thin layer of clothes to calculate the BMI according to the following equation for both groups (A&B):
  BMI = weight/height2 (kg/m2).
cortisol levels in blood | 12 weeks
  All women in both groups (A&B) will be evaluated before and after the treatment (12 weeks) to show serum cortisol level. A blood sample was taken from each female in both groups (A & B) before and after the treatment to measure the serum cortisol levels, which could reflect anxiety and pain intensity with decreased cortisol levels indicating decreased pain intensity. The cortisol level was assessed 5 days before the first day of the menstrual cycle preceding the treatment program and 5 days before the first day of the menstrual cycle at the end of treatment program,Blood sample of about 5 cm was drawn from the anticubital vein from all participants by disposable sterile syringe by vein puncture to determine plasma cortisol level. All blood samples were taken at 8-9 am and the norm cortisol level at 9 A.M ranges from 4.3-22.4 ug/dl.
Premenstrual syndrome score | 12 weeks
  The premenstrual syndrome scale comprised 40 questions with three sub-scales (Physiological, Psychological and Behavioural symptoms). This 5-point Likert- type scale consisting of 40 items. The measurements on the scale are set according to the following scoring system: the response Never was scored as "1", rarely as "2", sometimes as "3", very often as "4" and always as "5" points, the total score obtained from the sub-scales established the "PMSS total score." The scale's lowest score is 40 and highest score is 200. If the scale's total score reached 80 points or above, this indicates the occurrence of PMS. Increases in the scores indicate an increase in PMS severity.
Waist and hip circumference measurements | 12 weeks
  Waist circumference was measured at the narrowest point between xipho-sternum and the iliac crest at the end of a gentle expiration; hip circumference was measured at the maximum circumference at the level of femoral trochanter. Then, waist/hip ratio was calculated by dividing waist circumference on hip circumference. All measurements were taken for all patients in both groups (A&B), while the patient was in the standing position, before starting and after the end of the treatment course.

CONTACTS AND LOCATIONS:
Overall Officials: amal mo youseef, professor, Study Director — Cairo University
Locations (1):
- Yara Mostafa Soliman, Cairo, Egypt

REFERENCES:
- [Background] Quintana-Zinn FA, Whitcomb BW, Ronnenberg AG, Bigelow C, Houghton SC, Bertone-Johnson ER. Premenstrual Symptom Patterns and Behavioral Risk Factors in Young Women: A Cross-Sectional Study. J Womens Health (Larchmt). 2017 Oct;26(10):1099-1105. doi: 10.1089/jwh.2016.5921. Epub 2017 Jun 26. PMID 28650737
- [Background] Vaghela N, Mishra D, Sheth M, Dani VB. To compare the effects of aerobic exercise and yoga on Premenstrual syndrome. J Educ Health Promot. 2019 Oct 24;8:199. doi: 10.4103/jehp.jehp_50_19. eCollection 2019. PMID 31867375
- [Background] Itriyeva K. The effects of obesity on the menstrual cycle. Curr Probl Pediatr Adolesc Health Care. 2022 Aug;52(8):101241. doi: 10.1016/j.cppeds.2022.101241. Epub 2022 Jul 21. PMID 35871162